CLINICAL TRIAL: NCT01184222
Title: EFFICACY EVALUATION OF GREAT OCCIPITAL NERVE ELECTRICAL STIMULATION ON REBOUND HEADACHE AFTER WITHDRAWAL IN MEDICATION OVERUSE HEADACHE OCCURING IN MIGRAINE PATIENTS (SENGO-CAM Study)
Brief Title: Efficacy Evaluation Of Great Occipital Nerve Electrical Stimulation On Rebound Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 02-API-07
Record Dates: First submitted 2010-07-19; First posted 2010-08-18 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: HEADACHE
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm Active SENGO (Active Comparator): The patients will be hospitalised and managed by medication withdrawal and active GONS, surgically temporarily implanted.
  Interventions: Device: great occipital nerve stimulation
- Arm sham SENGO (Placebo Comparator): The patients will be hospitalised and managed by medication withdrawal and sham GONS, surgically temporarily implanted.
  Interventions: Device: great occipital nerve stimulation

INTERVENTIONS:
Device: great occipital nerve stimulation — * Active Comparator: Arm Active SENGO The patients will be hospitalised and managed by medication withdrawal and active GONS, surgically temporarily implanted.
  * Arm sham SENGO : The patients will be hospitalised and managed by medication withdrawal and sham GONS, surgically temporarily implanted.

SUMMARY:
SENGO-CAM study is a sham-controlled simple blind trial which aim is to study the efficacy of great occipital nerve stimulation (GONS) associated with medication withdrawal in the treatment of medication overuse headache occurring in migraine patients.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* migraine patient with medication overuse headache by non specific analgesics according to the ICHD-II diagnostic criteria
* failure of outpatient withdrawal
* Signature of informed consent.
* Affiliation to French national health and pensions organization

Exclusion Criteria:

* pregnancy (positive pregnancy test at pre-study) and breast-feeding
* patients with medication overuse headache by specific antimigraine treatment (triptans or/and ergot derivatives) according to the ICHD-II diagnostic criteria
* previous surgical treatment targeting great occipital nerves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Primary endpoint will be the comparison of the rate of headache-free patients, fourteen days after medication withdrawal, in both groups (GONS versus sham) | 14 days

SECONDARY OUTCOMES:
number of headache days during the 14 days withdrawal period | 14 days
maximal intensity and duration of rebound headache | 14 days
rescue medication used | 14 days
withdrawal facility perceived by the patient | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: FONTAINE Denys, PhD, Study Chair — Neurosurgery depatment - CHU Pasteur, Nice; LANTERI-MINET Michet, PhD, Study Chair — Neurosurgery department
Locations (4):
- France (4):
  - Neurology department - La timone, Marseille
  - Neurosurvery department, Nice
  - Headache Emergency Center, Paris
  - Neurology department - CHU Rangueil, Toulouse